CLINICAL TRIAL: NCT06882317
Title: A Study to Evaluate the Long Term Safety of CLBR001, a Lentiviral Based Chimeric Antigen Receptor, in Subjects Previously Administered CLBR001
Brief Title: Long Term Follow-up Study for Subjects Administered CLBR001
Status: Enrolling by invitation | Type: Observational
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Other Study IDs: CBR-CLBR001-3002
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Long Term Follow-Up
Keywords: Long Term Follow-Up (LTFU); CLBR001; Autologous Cell Therapy; Switchable CAR-T Cell; Cell and Gene Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen serum leftover following protocol-required testing of PK and ADA may be retained for future research or analytical development involving the same or related therapies or therapeutic areas, or for other relevant health research. This additional testing may involve genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLBR001 Treated Subjects: Subjects who received CLBR001 on any Calibr treatment study.
  Interventions: Other: Long Term Follow-Up

INTERVENTIONS:
Other: Long Term Follow-Up — No intervention is administered on this study. Subjects who have received CLBR001 autologous CAR-T cells in a primary Calibr treatment trial will be followed long term in line with FDA guidance.

SUMMARY:
The goal of this Long Term Follow-Up observational study is to monitor subjects who have received CLBR001, a lentiviral vector based chimeric antigen receptor, for delayed adverse events that may be associated with human gene therapies.

Participants will be followed for 15 years post-gene therapy administration date for safety and efficacy.

DETAILED DESCRIPTION:
In line with FDA guidance on Long Term Follow-Up (LTFU) after administration of human gene therapy products, any subject who receives CLBR001 on any Calibr treatment study will participate in LTFU on this study. Subjects will be enrolled following completion on the applicable treatment study and followed for 15 years post-CLBR001 administration in order to assess the long term safety of CLBR001.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received at least one CLBR001 cell dose.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received CLBR001.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2044-02 (Estimated); Study Completion 2044-02 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events as assessed by CTCAE v5.0. | To 15 years post-CLBR001 administration.
  To assess the long term safety of CLBR001 in subjects by evaluating the incidence, duration, and outcome of adverse events (including adverse events of special interest, CLBR001-related adverse events and serious adverse events), as assessed by CTCAE v5.0.
Number of subjects with replication competent lentivirus (RCL). | To 15 years post-CLBR001 administration.
  To assess the long term safety of CLBR001 in subjects by evaluating the proportion of subjects with detectable RCL from CLBR001.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Calibr-Skaggs Institute for Innovative Medicines
Locations (1):
- Virtual Research Group- Premier Research, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No